CLINICAL TRIAL: NCT02760745
Title: Fever and Shivering: Frequency Among Children Visiting the Emergency Department and Its Role in Predicting Serious Bacterial Infection
Brief Title: Fever and Shivering: Frequency and Role in Predicting Serious Bacterial Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Assaf Harofeh MC, Director Pediatric Emergency Unit, Assaf-Harofeh Medical Center
Other Study IDs: ASF-0207-15
Record Dates: First submitted 2016-03-24; First posted 2016-05-04 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Febrile Shivering; Severe Bacterial Infection
Keywords: fever; shivering; chills; rigors; severe bacterial infection
MeSH Terms: conditions — Bacterial Infections; Fever; Chills

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood, urine, stool, csf, throat culture, joint fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Febrile Shivering
  Interventions: Other: Ancillary tests
- Fever without Shivering
  Interventions: Other: Ancillary tests

INTERVENTIONS:
Other: Ancillary tests — Blood culture, complete blood count, crp, urinalysis for all patients. If clinically indicated: Urine culture, chest x ray, csf culture, stool culture, joint fluid culture

SUMMARY:
Febrile shivering in the pediatric population is assumed to be related to a Severe Bacterial Infection (SBI). Research supporting this assumption is scant. The purpose of this study is to describe the frequency of febrile shivering in the pediatric population arriving at the emergency department and to define its role in predicting a SBI.

DETAILED DESCRIPTION:
Background: Fever is a common complaint and lacking localizing signs poses a diagnostic dilemma, mostly, but not only, in children under 3 years of age. Recent years studies found common clinical markers for a Serious Bacterial Infection (SBI) to be ineffective in confirming or ruling out a suspected SBI in an environment with low prevalence of SBI such as developed countries. Shivering (chills, rigors) during a febrile illness is a common complaint in children but it's true incidence is unknown. It is assumed that shivering appears more frequently in children with SBI but only one study in the pediatric population was found to support this assumption. No studies were found to describe the frequency of shivering in the emergency department. Study purpose: To describe the frequency of febrile shivering in the pediatric population arriving at the emergency department and it's relation to a Severe Bacterial Infection. Participants: Children in the age range of 3 months to 18 years presenting with fever. Intervention: During the study time frame the frequency of febrile shivering will be documented . Patients with febrile shivering who meet the inclusion criteria, a sepsis workup will be done including blood samples for inflammatory markers, blood culture, urinalysis and urine culture when a urinary tact infection is suspected. Other systems (CSF sampling, joint fluid aspiration, stool culture, chest x ray) will be examined according to an appropriate history and clinical suspicion. The same work up will be done in next consecutive patient presenting with fever without shivering. Results: The frequency of febrile shivering, positive cultures, lobar pneumonia in a chest x ray. A comparison between the study and the control group will be made. Categorical variables will be compared using the Chi square test or Fisher exact test (as appropriate). Continuous variables will be compared using the student t test or Mann Whitney test. The relation between a bacterial infection and clinical variables will be analyzed using a logistic regression. Study group size: This is a pilot study. Investigators will use a convenience sample of all children admitted with shivering during the study period.

Safety: All examinations will be held by the emergency department organic staff in the same routine methods done otherwise outside the study settings. The emergency department and hospital protocols for patients identification and infection control will be carried out before invasive procedures. Ethics: Parents will be asked for their agreement to answer a questioner as part of the study and their agreement will be documented. Informed consent will be asked for each patient, of the legal guardian. The study will be held according to the ethics rules of the Helsinki declaration and was approved by the local Ethics board. Access to the database will be restricted to the study investigators. The database will be encrypted by a password. After gathering the data and before statistical analysis information identifying the patients will be removed. The importance of the study: Fever in children is a common complaint frequently posing a dilemma on the extent of workup needed beyond clinical evaluation. This study aims to examine the frequency of shivering among children presenting to the ED with fever , its ability to predict the risk of severe bacterial infection.

ELIGIBILITY:
Inclusion Criteria:

* fever at least during the last day
* shivering during current febrile illness
* no shivering during current febrile illness if recruited to the control group Exclusion Criteria: (for cases and controls)
* immune deficiency
* antibiotics treatment up to 48 hours before the presentation
* presentation following febrile convulsion
* non Hebrew speaking guardians

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients arriving at the pediatric emergency department with fever
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of febrile children who experienced shivering | Within 7 days from the beginning of fever
  Proportion of febrile children who experienced shivering
Severe bacterial infection | Within 7 days from enrollment
  positive blood cultures (not including common skin pathogens / contaminants), Positive urine culture, Positive csf culture, Alveolar Infiltrate on CXR, positive joint fluid culture.
  The number of patients who had at least one positive result in the above mentioned parameters.

SECONDARY OUTCOMES:
High inflammatory markers | Within 24 hours of enrollment
  The number of patients who had CRP higher than twice the normal range or WBC higher than 15,000.
Antibiotics Treatment | Within 24 hours of enrollment
  number of patients treated with antibiotics
hospitalization | Within 24 hours of enrollment
  number of patients admitted to the hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf Harofeh MC, Ẕerifin, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Baraff LJ. Management of infants and young children with fever without source. Pediatr Ann. 2008 Oct;37(10):673-9. doi: 10.3928/00904481-20081001-01. PMID 18972849
- [Background] McCarthy PL, Sharpe MR, Spiesel SZ, Dolan TF, Forsyth BW, DeWitt TG, Fink HD, Baron MA, Cicchetti DV. Observation scales to identify serious illness in febrile children. Pediatrics. 1982 Nov;70(5):802-9. No abstract available. PMID 7133831
- [Background] Brauner M, Goldman M, Kozer E. Extreme leucocytosis and the risk of serious bacterial infections in febrile children. Arch Dis Child. 2010 Mar;95(3):209-12. doi: 10.1136/adc.2009.170969. PMID 20308337
- [Background] Van den Bruel A, Haj-Hassan T, Thompson M, Buntinx F, Mant D; European Research Network on Recognising Serious Infection investigators. Diagnostic value of clinical features at presentation to identify serious infection in children in developed countries: a systematic review. Lancet. 2010 Mar 6;375(9717):834-45. doi: 10.1016/S0140-6736(09)62000-6. Epub 2010 Feb 2. PMID 20132979
- [Background] Craig JC, Williams GJ, Jones M, Codarini M, Macaskill P, Hayen A, Irwig L, Fitzgerald DA, Isaacs D, McCaskill M. The accuracy of clinical symptoms and signs for the diagnosis of serious bacterial infection in young febrile children: prospective cohort study of 15 781 febrile illnesses. BMJ. 2010 Apr 20;340:c1594. doi: 10.1136/bmj.c1594. PMID 20406860
- [Background] Richardson M, Lakhanpaul M; Guideline Development Group and the Technical Team. Assessment and initial management of feverish illness in children younger than 5 years: summary of NICE guidance. BMJ. 2007 Jun 2;334(7604):1163-4. doi: 10.1136/bmj.39218.495255.AE. No abstract available. PMID 17540946
- [Background] Tal Y, Even L, Kugelman A, Hardoff D, Srugo I, Jaffe M. The clinical significance of rigors in febrile children. Eur J Pediatr. 1997 Jun;156(6):457-9. doi: 10.1007/s004310050638. PMID 9208242
- [Background] Lee CC, Wu CJ, Chi CH, Lee NY, Chen PL, Lee HC, Chang CM, Ko NY, Ko WC. Prediction of community-onset bacteremia among febrile adults visiting an emergency department: rigor matters. Diagn Microbiol Infect Dis. 2012 Jun;73(2):168-73. doi: 10.1016/j.diagmicrobio.2012.02.009. Epub 2012 Mar 29. PMID 22463870